CLINICAL TRIAL: NCT00719199
Title: Open-label Phase 1b Study of FOLFIRI Plus Cetuximab Plus IMO-2055 in Patients With Colorectal Cancer Who Have Progressed Following Chemotherapy for Advanced or Metastatic Disease
Brief Title: Study of FOLFIRI Plus Cetuximab Plus IMO-2055 in Patients With Colorectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor will discontinue further development of EMD 1201081
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMO-2055-210; EMR200068_210
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; metastatic cancer; prior therapy; 1b
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — IMO-2055; Cetuximab; IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): IMO 2055 is a novel phosphorothioate oligodeoxynucleotide that is an agonist of Toll-like Receptor 9 (TLR9).
  Interventions: Drug: IMO-2055; Drug: Cetuximab; Drug: FOLFIRI

INTERVENTIONS:
Drug: IMO-2055 — SC weekly injections
Drug: Cetuximab — given weekly through intravenous administration. Cycle 1 Day 1 dose given at 400mg/m2, all subsequent doses given at 250 mg/m2.
Drug: FOLFIRI — Given day 1 of each cycle

SUMMARY:
Open-label phase 1b trial. Study treatment will be administered in 3 week cycles.

There are two distinct parts in this study:

* Part 1: Dose escalation from IMO-2055
* Part 2: Once a recommended phase 2 dose is found additional tolerability and pharmacodynamics will be explored

DETAILED DESCRIPTION:
* Part 1: Dose escalation of IMO-2055, including 3 dose groups. Once a recommended phase 2 dosage (RP2D) of IMO-2055 given concomitantly with FOLFIRI and cetuximab is found the selected cohort will be expanded by an additional 6 to 9 patients (to a total of 12 patients) for confirmation of the RP2D and combination treatment regimen.
* Part 2: A final cohort of 12 patients (Cohort 6) will be enrolled simultaneously to explore tolerability and pharmacodynamics in patients treated with the RP2D of IMO-2055 in combination with FOLFIRI with cetuximab.

ELIGIBILITY:
Inclusion Criteria:

Patients must satisfy all the following inclusion criteria in order to be eligible for the study:

1. Signed written informed consent prior to any study-specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.
2. Male or female patients aged ≥ 18 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Histologically confirmed adenocarcinoma of the colon or rectum with advanced or metastatic disease.
5. Patients whose disease has recurred or progressed during or after completion of at least one (1) standard regimen of cytotoxic agents. Patients may have had any number of prior regimens as long as the other entry criteria are met. Preferred patients are those who have progressed on first line FOLFIRI or FOLFOX with or without bevacizumab. Patients may have had prior exposure to monoclonal antibodies such as cetuximab, bevacizumab or panitumumab.
6. All clinically significant adverse events of any prior chemotherapy, surgery or radiotherapy must have resolved to CTCAE v3.0 grade ≤ 1. Neuropathy of CTCAE v3.0 grade ≤ 2 will be allowed but the neuropathy should be closely monitored throughout the trial.
7. A minimum of 4 weeks must occur between last receipt of chemotherapy, biotherapy, radiotherapy, or major surgery and registration.
8. Be willing and able to comply with the protocol for the duration of the study.
9. If prior malignancy was diagnosed, other than colorectal, no evidence of disease from that cancer, off all therapy for that cancer and recovered to grade 1 or less toxicity from prior treatment.

Exclusion Criteria:

Patients with any of the following will be excluded from participation in the study:

Disease

1. Known central nervous system (CNS) metastases unless controlled for ≥ 4 months without the use of steroids.
2. Patients who are candidates for neoadjuvant "conversion" therapy followed by curative surgery.

   Prior Treatments
3. Prior pelvic irradiation.
4. Administration of any investigational agent (therapeutic or diagnostic), within 4 weeks prior to first study dosing.
5. Patients with a prior history of cetuximab hypersensitivity may be admitted to Part 1 of the study only.

   Other Concomitant Medications
6. Chronic oral or intravenous corticosteroids. (Note: Doses ≤ 5 mg/day of prednisone or equivalent are permitted. Topical, inhaled and intra-articular corticosteroids are allowed.)
7. Therapeutic anticoagulation (warfarin > 1 mg/day or heparin). Low-dose warfarin for port prophylaxis and low-molecular weight heparin at therapeutic doses are allowed.

   Laboratory
8. The following laboratory results:

   * Hemoglobin < 9.0 g/dL Absolute neutrophil count < 1.5 x 109/L Platelet count < 100 x 109/L
   * Total bilirubin > 1.5 x upper limit of normal (ULN)
   * ALT or AST > 2.5 x ULN (> 5 x ULN if liver metastases present)
   * Alkaline phosphatase > 2.5 x ULN (> 5 x ULN if liver metastases present, or > 10 x ULN in case of the presence of bone metastases)
   * Serum creatinine > 1.5 x ULN
   * Albumin < 2.5 g/dL Other Conditions or Procedures
9. Grade 3 or 4 non-hematological toxicity or febrile neutropenia related to previous irinotecan-based regimens.
10. Homozygous for the UGT1A1*28 allele.
11. Known hypersensitivity to murine proteins or oligonucleotides.
12. Pregnant or breast-feeding women.
13. Women of childbearing potential with either positive or no pregnancy test at baseline. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential.
14. Men or women of childbearing potential who refuse or who are unable to use an acceptable means of contraception during the study.
15. History of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the Investigator to be clinically significant precluding informed consent or interfering with compliance.
16. Pre existing autoimmune or antibody-mediated diseases, including, but not limited to, the following: organ allografts, systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome and autoimmune thrombocytopenia, known Gilbert's syndrome.
17. Signs/symptoms of bowel obstruction or pseudo-obstruction or history of inflammatory bowel disease.
18. Clinically significant (i.e., active) cardiac disease (e.g., congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 6 months.
19. Interstitial pneumonia or extensive symptomatic fibrosis of the lungs.
20. Serious uncontrolled concomitant disease, intercurrent infections, or other known medical conditions that in the opinion of the Investigator puts the patient at increased risk for significant toxicities from treatment, such as hypertension, uncontrolled by medication, chronic hepatitis (viral or other) or cirrhosis, known human immunodeficiency virus (HIV) infection, or uncontrolled diabetes.
21. Legal incapacity or limited legal capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-01; Primary Completion 2011-04 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
• The primary objective of this study is to determine the recommended phase 2 dose of IMO 2055 when combined with FOLFIRI and cetuximab in patients with histologically proven advanced or metastatic colorectal cancer (CRC). | 10 months from first patient in, Oct 2010

SECONDARY OUTCOMES:
• To evaluate the safety of weekly IMO 2055 combined with FOLFIRI plus cetuximab. | Assessed weekly at patient visits
• To investigate the pharmacokinetics (PK) of IMO-2055. | Assessed weekly at patient visits until Cycle 4
• To investigate the tolerability and pharmacodynamic (PD) effects of dexamethasone scheduling with IMO 2055 and FOLFIRI. | Assessed weekly at patient visits until Cycle 4
• To investigate potential signs of efficacy using the Response Evaluation Criteria for Solid Tumors (RECIST) response rate in patients with measurable disease. | Every six weeks
• To investigate progression-free survival (PFS) and overall survival for up to one year in all patients. | Every three months
• To investigate results of subsequent therapy (if any) in all patients. | Every three months
• To investigate potential markers of IMO 2055 immune activation and effect on cellular immunity. | Assessed weekly at patient visits until Cycle 4

CONTACTS AND LOCATIONS:
Overall Officials: Phil Breitfeld, MD, Study Director — EMD Serono
Locations (5):
- United States (5):
  - Georgetown University Lombardi Cancer Center, Washington D.C., District of Columbia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Cancer Therapy & Research Center, San Antonio, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas

REFERENCES:
- [Derived] Chan E, Kwak EL, Hwang J, Heiskala M, de La Bourdonnaye G, Mita M. Open-label phase 1b study of FOLFIRI plus cetuximab plus IMO-2055 in patients with colorectal cancer who have progressed following chemotherapy for advanced or metastatic disease. Cancer Chemother Pharmacol. 2015 Apr;75(4):701-9. doi: 10.1007/s00280-015-2682-2. Epub 2015 Jan 28. PMID 25627002